CLINICAL TRIAL: NCT05609864
Title: Drug Wastage : Observational Study in the Operating Rooms of France
Acronym: GAME-OvBLOC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Sainte-Anne Military Teaching Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-CHITS-001
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Drug Use
Keywords: Drug wastage; Green Anesthesia; Environmental sustainability; Injectable drugs; Eco-design of care; Operating Room

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Injectable drugs: Patient's data and data relating to prepared/administrated/discarded injectable drugs will be collected during 24 hours in the operating rooms by anesthesia department
  Interventions: Other: Quantification of injectable drugs wastage

INTERVENTIONS:
Other: Quantification of injectable drugs wastage — Drugs are prescribed at discretion of physicians. For each patient who have anesthesia in the operating room, all labelled syringes having contained drugs (name + dilution) are collected and analyzed.

SUMMARY:
Environmental awareness is leading medical field to question its responsibility and possibilities for action.

Drug residues can have a major environmental impact as per their bioaccumulation, toxicity and persistence characteristics, depending on where they are discarded. In France, drug residues should be disposed of by incineration, but in practice this is not systematic. Moreover, data on drug wastage in the operating rooms by anesthesia department are rare.

The GAME-OvBLOC observational study aim to evaluate drug wastage in the operating rooms by anesthesia department in France and to propose ways of improving health care practices.

DETAILED DESCRIPTION:
Observational study with data collection over a 24-hour business day. Data collected refer to healthcare team's practices and patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will need an anesthesia act in operating room during a 24 hours period

Exclusion Criteria:

* Patient opposition to participate in the study or parents opposition if the patient is a child or patient family opposition if the patient is not capable of being informed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who will need an anesthesia act in operating room during a 24 hours period
Sampling Method: Non-Probability Sample
Enrollment: 3763 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Ratio of overall wastage in milliliter (mL) of prepared and discarded injectable drugs, to overall volume in milliliter (mL) of prepared injectable drugs | 24 hours
  Wastage is defined as : any prepared and unused drug that remains in syringe

SECONDARY OUTCOMES:
Reason for discarding drug residues | 24 hours
  The reason of waste full syringe will be noticed : 1/ prepared in advance and not used ; 2/ prescription change ; 3/ preparation error ; 4/ other reason
Describe drug wastage for each kind of surgery/anesthesia | 24 hours
  Drug wastage according to type of surgery and anaesthesia
Drug residues discarding process | 24 hours
  Questionnaire on nursing practices on the choice of waste disposal circuits according to drugs
Cost of overall injectable drugs wastage | 24 hours
  Estimated cost of drug residues will be evaluated for each drug by the following formula :
  volume of discarded injectable drugs x theoretical price
Describe drug wastage for each age group | 24 hours
  Drug wastage according to the following age groups : adult (≥18 years old) and pediatrics (< 1 year old, 1-5 years old, ≥ 6 years old)
Describe waste and environmental impact of used plastic syringes | 24 hours
  Number and volume of used syringes, use of pre-filled syringes, refilling of syringes and multi-patient use.
  Environmental impact is indirectly assessed by type of plastic used and the transport distance from the production site to France.
Use of alternative to injectable drugs | 24 hours
  Alternatives : local anaesthesia and anaesthetic gases

CONTACTS AND LOCATIONS:
Overall Officials: Erwan D'Aranda, MD, Study Director — Sainte-Anne Military Teaching Hospital (Hôpital d'instruction des armées Sainte Anne)
Locations (83):
- France (80):
  - Centre Hospitalier de Cannes, Cannes, Alpes-Maritimes
  - Centre Hospitalier de Charleville-Mézières, Charleville-Mézières, Ardennes
  - Centre Hospitalier Jacques Puel, Rodez, Aveyron
  - CHU de Strasbourg - IHU, Strasbourg, Bas-Rhin
  - Hôpital La Timone (AP-HM), Marseille, Bouches-du-Rhône
  - Hôpital Nord (AP-HM), Marseille, Bouches-du-Rhône
  - CHU de Caen, Caen, Calvados
  - Centre Hospitalier Henri Mondor, Aurillac, Cantal
  - Groupe Hospitalier Littoral Atlantique, La Rochelle, Charente-Maritime
  - Centre Hospitalier de Brive-la-Gaillarde, Brive-la-Gaillarde, Corrèze
  - CHU de Dijon, Dijon, Côte d'Or
  - CHU Jean Minjoz, Besançon, Doubs
  - Centre Hospitalier de Valence, Valence, Drôme
  - Centre hospitalier Sud Francilien, Corbeil-Essonnes, Essonne
  - HIA Clermont Tonnerre, Brest, Finistère
  - CHRU de Brest, Brest, Finistère
  - Centre Hospitalier de Cornouailles, Quimper, Finistère
  - CHU de Nîmes, Nîmes, Gard
  - CHU de Bordeaux - Groupe hospitalier Pellegrin, Bordeaux, Gironde
  - Centre Hospitalier d'Arcachon, La Teste-de-Buch, Gironde
  - CHU de Bordeaux, Groupe Sud, Pessac, Gironde
  - Clinique mutualiste de Pessac, Pessac, Gironde
  - CHU de Limoges, Limoges, Haute Vienne
  - Clinique des Cèdres, Cornebarrieu, Haute-Garonne
  - Clinique la Croix du Sud, Quint-Fonsegrives, Haute-Garonne
  - Clinique de l'Union, Saint-Jean, Haute-Garonne
  - CHU de Toulouse - Hôpital Rangueil, Toulouse, Haute-Garonne
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay, Haute-Loire
  - HIA Percy Clamart, Clamart, Hauts-de-Seine
  - Hôpital Marie Lannelongue, Le Plessis-Robinson, Hauts-de-Seine
  - CHU de Rennes - Pontchaillou, Rennes, Ille-et-Vilaine
  - CHU de Rennes - Hôpital Sud, Rennes, Ille-et-Vilaine
  - Clinique mutualiste La Sagesse, Rennes, Ille-et-Vilaine
  - CHU de Grenoble, Grenoble, Isère
  - CHU de la Réunion, Saint-Denis, La Réunion
  - Centre Hospitalier de Dax, Dax, Landes
  - Centre Hospitalier de l'Agglomération Montargoise, Amilly, Loiret
  - Clinique de l'Archette, Olivet, Loiret
  - CHU d'Angers, Angers, Maine-et-Loire
  - Institut Godinot, Reims, Marne
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Groupe Hospitalier Bretagne Sud, Lorient, Morbihan
  - Centre Oscar Lambret, Lille, Nord
  - CHU de Lille - Institut coeur poumon, Lille, Nord
  - CHU de Lille - Hôpital Huriez, Lille, Nord
  - CHU de Lille - Hôpital Jeanne de Flandre, Lille, Nord
  - CHU de Lille - Hôpital Roger Salengro, Lille, Nord
  - Hôpital privé Arras les Bonnettes, Arras, Pas-de-Calais
  - Centre Hospitalier de Lens, Lens, Pas-de-Calais
  - CHU de Clermont-Ferrand, Clermont-Ferrand, Puy-de-Dôme
  - Clinique de la Plaine Santé, Clermont-Ferrand, Puy-de-Dôme
  - Clinique Aguilera, Biarritz, Pyrénées-Atlantiques
  - Centre Hospitalier de Pau, Pau, Pyrénées-Atlantiques
  - Hôpital mère-enfant (HCL), Bron, Rhône
  - Hôpital Edouard Herriot, Lyon, Rhône
  - Centre Léon Bérard, Lyon, Rhône
  - Clinique de la Sauvegarde, Lyon, Rhône
  - CHU de Rouen, Rouen, Seine-Maritime
  - CHU d'Amiens, Amiens, Somme
  - Clinique Victor Pauchet, Amiens, Somme
  - Centre Hospitalier Intercommunal Castres-Mazamet, Castres, Tarn
  - Hôpital Nord Franche-Comté, Trévenans, Territoire De Belfort
  - Hôpital Privé de la Chataigneraie, Beaumont, Val d'Oise
  - Hôpital NOVO - Site de Beaumont-sur-Oise, Beaumont-sur-Oise, Val d'Oise
  - Hôpital NOVO - Site de Pontoise, Cergy-Pontoise, Val d'Oise
  - Institut Gustave Roussy, Villejuif, Val-de-Marne
  - Centre Hospitalier Intercommunal de Villeneuve Saint Georges, Villeneuve-Saint-Georges, Val-de-Marne
  - Sainte-Anne Military Teaching Hospital, Toulon, Var
  - Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer, Toulon, Var
  - Hôpital Robert Schuman-Groupe UNEOS, Vantoux, Vaucluse
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon, Vendée
  - Hôpital Lariboisière (AP-HP), Paris
  - Hôpital Saint Louis (AP-HP), Paris
  - Hôpital Trousseau (AP-HP), Paris
  - Hôpital La Pitié-Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hôpital Tenon (AP-HP), Paris
  - Institut mutualiste Montsouris, Paris
  - Hôpital Paul Brousse (AP-HP), Villejuif
- CHU de Guadeloupe, Pointe-à-Pitre, Guadeloupe
- Centre Hospitalier de Mayotte, Mamoudzou, Mayotte
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGain F, Muret J, Lawson C, Sherman JD. Environmental sustainability in anaesthesia and critical care. Br J Anaesth. 2020 Nov;125(5):680-692. doi: 10.1016/j.bja.2020.06.055. Epub 2020 Aug 12. PMID 32798068
- [Background] Barbariol F, Deana C, Lucchese F, Cataldi G, Bassi F, Bove T, Vetrugno L, De Monte A. Evaluation of Drug Wastage in the Operating Rooms and Intensive Care Units of a Regional Health Service. Anesth Analg. 2021 May 1;132(5):1450-1456. doi: 10.1213/ANE.0000000000005457. PMID 33667211
- [Background] Mankes RF. Propofol wastage in anesthesia. Anesth Analg. 2012 May;114(5):1091-2. doi: 10.1213/ANE.0b013e31824ea491. Epub 2012 Mar 13. PMID 22415537
- [Background] Ramstrom H, Martini S, Borgendahl J, Agerstrand M, Larfars G, Ovesjo ML. Pharmaceuticals and Environment: a web-based decision support for considering environmental aspects of medicines in use. Eur J Clin Pharmacol. 2020 Aug;76(8):1151-1160. doi: 10.1007/s00228-020-02885-1. Epub 2020 May 9. PMID 32388641
- See also: Direction générale de la santé. Pour Une Bonne Gestion Des Déchets Produits Par Les Établissements de Santé et Médico-Sociaux. Déchets Issus de Médicaments. Déchets Liquides. Ministère des Affaires sociales et de la Santé; 2016. — https://solidarites-sante.gouv.fr/IMG/pdf/pour_une_bonne_gestion_des_dechets_produits_par_les_etablissements_de_sante_et_medico-sociaux.pdf